CLINICAL TRIAL: NCT06675708
Title: Study of the Effectiveness of Creatine on Pain, Fatigue, and Muscle Architectural Variables in Patients Witg Fibromyalgia.
Brief Title: Effectiveness of Creatine on Pain, Fatigue, and Muscle Architectural Variables in Patients Witg Fibromyalgia.
Acronym: SECPFMAPFM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Edurne Úbeda D'Ocasar, Doctor Edurne Úbeda D'Ocasar, Camilo Jose Cela University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FIBYSAR2
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
Keywords: Creatine; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Creatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The creatine experimental group will receive 20g of creatine for 5 days, divided into 4 equal doses, followed by 5g/day as a single dose for the duration of the trial.
  Interventions: Dietary Supplement: Creatine
- Placebo group (Placebo Comparator): The placebo group will receive 20g of dextrose for 5 days, divided into 4 equal doses, followed by 5g/day as a single dose for the duration of the trial
  Interventions: Dietary Supplement: Dextrose

INTERVENTIONS:
Dietary Supplement: Creatine — From the total sample obtained after recruitment, randomization will be performed using the SPSS statistical program, creating two groups. One experimental group will receive creatine supplementation, and the other group will receive a placebo through dextrose administration. In both cases, the doses will be administered in the same manner to both groups
  Arms: Experimental group
Dietary Supplement: Dextrose — From the total sample obtained after recruitment, randomization will be performed using the SPSS statistical program, creating two groups. Dextrose group will be administered in the same manner as creatine to the experimental group. The doses will be prepared in the same way for both groups.
  Arms: Placebo group

SUMMARY:
Creatine, a non-protein organic amino acid, is synthesized from arginine, glycine, and methionine. The use of creatine has been shown to be effective in healthy subjects, providing benefits primarily in terms of strength, which has been the main factor studied. In patients with various conditions, including pain, creatine supplementation has demonstrated a reduction in pain and even cognitive improvements.

Due to creatine's general improvement in muscular endurance and fatigue.

DETAILED DESCRIPTION:
Through this study, we aim to analyze whether creatine supplementation can be beneficial in reducing symptoms in patients with Fibromyalgia. Previous studies have demonstrated its benefits, and therefore, we want to evaluate if these benefits can manifest in a shorter time compared to previous studies in patients with Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FM
* aged between 18 and 75 years
* agree to participate and sign the informed consent

Exclusion Criteria:

* who do not have recent surgeries
* patients with reduced mobility
* adequate level of comprehension to be able to answer the questionnaires that will be provided in the study
* If they are taking antihypertensive medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Algometer | baseline; after finishing the treatment (two months)
  Algometer points: Using an algometer, the pain threshold at each tender point is measured in kg/cm. The higher the value obtained, the less pain the subject has.
VAS | baseline; after finishing the treatment (two months)
  Visual Analogic Scale: this self-referenced scale ranges from 0 to 10 where 0 is no pain at all and 10 indicates the worst possible pain endured. The higher the score, the greater the pain
Circometry | baseline; after finishing the treatment (two months)
  Contour measurements: The contour of the segment selected for the study will be measured using a tape measure. It is measured in centimeters. the greater the number of centimeters, the greater the diameter and therefore the worse the condition or greater the liquid retention of the subject.
Dynamometer | baseline; after finishing the treatment (two months)
  upper limb grip strength: this measuring tool measures upper limb grip strength. the higher the value, the better the subject's state of strength
Chair test | baseline; after finishing the treatment (two months)
  number of squats for 30 seconds: this test consists of seeing how many squats can be done in the test time. The greater the number of squats, the better the subject will be.
Timed up and go | baseline; after finishing the treatment (two months)
  balance test: The Timed Up and Go Test is an easy-to-use test to assess the risk of falls.The shorter the test time, the lower the risk of falling.
anthropometric measurements | baseline; after finishing the treatment (two months)
  anthropometric measurements with the uso of the Tanita
muscular architectural stockings | baseline; after finishing the treatment (two months)
  taking architectural muscle averages using an ultrasound scanner
Pittsburgh | baseline; after finishing the treatment (two months)
  sleep quality questionnaire: This test has values from 0 to 21 points maximum. It is interpreted that the higher the score, the worse the quality of sleep.
FIQ | baseline; after finishing the treatment (two months)
  fibromyalgia impact questionnaire: The total FIQ score is between 0-100 as each of the items has a score of 0-10 once adapted. Thus, 0 represents the highest functional capacity and quality of life and 100 the worst state.
SARC-F | baseline; after finishing the treatment (two months)
  questionnaire to measure sarcopenia risk: The SARC-F is a quick and easy instrument for detecting the risk of sarcopenia, which asks the degree of difficulty an older adult has in performing 4 functional activities. A score greater than 4 indicates risk of sarcopenia.
HADS | baseline; after finishing the treatment (two months)
  to evaluate emotional distress in patients with different chronic conditions, assessing cognitive and behavioral symptoms of anxiety and depression. The HADS is composed of two subscales: Depression and Anxiety, each with seven items. The score of each subscale can vary between 0 and 21, since each item presents four response options, ranging from absence/minimal presence = 0, to maximum presence = 3.

SECONDARY OUTCOMES:
socio-demographic variables | baseline
  socio-demographic variables (age, weight, height, medication intake, marital status, employment status, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Úbeda-D'Ocasar, Doctor, Principal Investigator — University Camilo José Cela
Locations (1):
- University Camilo José Cela, Madrid, Spain